CLINICAL TRIAL: NCT06510673
Title: Extracorporeal Shock Wave Therapy Versus High Power LASER Therapy for the Treatment of Females With Calcaneal Spur
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Suez University (Other); Badr University (Other); Helwan University (Other)
Responsible Party: Principal Investigator, Mina Magdy Wahba, Lecturer, Suez University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SU1
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Calcaneal Spur
MeSH Terms: conditions — Heel Spur | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Shockwave therapy (Experimental): Shockwave therapy for calcaneal spur
  Interventions: Other: Shockwave therapy
- High-power LASER therapy (Experimental): High-power LASER therapy for calcaneal spur
  Interventions: Other: High power LASER
- Control (Sham Comparator): cold application with receive 6 sessions of sham LASER therapy.
  Interventions: Other: Ice application; Other: Sham LASER
- Platelet rich plasma (Experimental): Platelet-rich plasma injection for the heel
  Interventions: Drug: Platelet rich plasma

INTERVENTIONS:
Drug: Platelet rich plasma — Platelet-rich plasma for the heel
  Arms: Platelet rich plasma
Other: High power LASER — High power LASER sessions for the heel
  Arms: High-power LASER therapy
Other: Shockwave therapy — Shockwave therapy sessions for the heel
  Arms: Shockwave therapy
Other: Ice application — Ice application for the heel
  Arms: Control
Other: Sham LASER — Sham LASER for the heel
  Arms: Control

SUMMARY:
PURPOSE: To compare the effect of Extracorporeal shock wave therapy and high-power LASER therapy for the treatment of patients with calcaneal spur Background: Calcaneal spur is a common musculoskeletal disorder of the foot that affect the quality-of-life Conservative treatment modalities include, cold application, platelet-rich plasma therapy (PRP), shoe modification, therapeutic ultrasound, extracorporeal shock wave therapy (ESWT), laser therapy (LLLT) are commonly used in the treatment of calcaneal spur.

HYPOTHESES: There will be difference between Extracorporeal shock wave therapy and High- power LASER therapy on pain intensity in patients with calcaneal spur There will be difference between Extracorporeal shock wave therapy and High- power LASER therapy on function in patients with calcaneal spur. There will be difference between Extracorporeal shock wave therapy and High- power LASER therapy on the size of calcaneal spur in patients with calcaneal spur.

RESEARCH QUESTION: Is there any difference between the effect of Extracorporeal shock wave therapy and High-power LASER on calcaneal spur?

ELIGIBILITY:
Inclusion Criteria:

diagnosed with calcaneal spur based on clinical examination and radiological findings.

Exclusion Criteria:

were as follows: acute trauma to the foot, history of fracture or surgery, lower extremity neurological deficit, polyneuropathy, radicular pain, autoimmune diseases tumor, thrombosis, soft tissue or bone infection, or skin disorder.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain Visual Analog Scale | Baseline and after one month
  It is a self reported outcome which is a 10 cm line with zero at one end indicating no pain and 10 at the other end indicating maximum pain. Patient will be asked to mark the current pain on the scale and the distance from the starting point (0) will be measured
foot function index. | Baseline and after one month
  measure the impact of foot pathology on function in terms of pain, disability and activity restriction. it is a self-administered index
calcaneal Spur length | Baseline and after one month
  Spur length will be measured by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Elsayed, Study Chair — Department of Physical therapy for Woman's Health, Faculty of Physical Therapy, Badr University in Cairo, Cairo, Egypt; Doha Hamed, Study Chair — Basic Sciences Department, Faculty of Physical Therapy, Badr University in Cairo; Ahmed Zakaria, Study Chair — Department of orthopedic surgery, Helwan University; Omnya Samy, Study Director — Department of Physical Therapy for Pediatrics and Pediatric Surgery, Faculty of Physical Therapy, Badr University in Cairo; Fatma Zidan, Study Director — Department of Physical therapy for Neuromuscular Disorders & its Surgery, Faculty of Physical Therapy, Badr University in Cairo; Doaa Saeed, Study Chair — Department of Physical Therapy for Women's Health, Faculty of Physical Therapy, Badr University in Cairo, Cairo, Egypt
Locations (1):
- Badr University in Cairo (BUC), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No